CLINICAL TRIAL: NCT04084444
Title: Efficacy and Safety of T8 on Treating Chronic Abnormal Immune Activation in HIV/AIDS Patients: A Multicenter, Randomized, Double-blind, Dose-finding, Placebo-controlled Study
Brief Title: Safety and Efficacy of T8 on Treating Chronic Abnormal Immune Activation in HIV/AIDS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T8-201
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-07

CONDITIONS: Chronic Abnormal Immune Activation in HIV/AIDS
Keywords: Chronic abnormal immune activation; AIDS; T8; Efficacy; Safety
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T8 tablet 0.5mg (Experimental): Oral T8 tablet with HARRT, 0.5mg, once daily for 48 week
  Interventions: Drug: T8 tablet 0.5mg
- T8 tablet 1mg (Experimental): Oral T8 tablet with HARRT, 1mg, once daily for 48 week
  Interventions: Drug: T8 tablet 1mg
- Placebo (Placebo Comparator): Oral Placebo with HARRT, once daily for 48 week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: T8 tablet 0.5mg — Immune regulation, inhibition of acute nonspecific inflammation and chronic inflammation.
  Other Names: Leiteng Shu
  Arms: T8 tablet 0.5mg
Drug: T8 tablet 1mg — Immune regulation, inhibition of acute nonspecific inflammation and chronic inflammation.
  Other Names: Leiteng Shu
  Arms: T8 tablet 1mg
Drug: Placebo — Blank control.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, dose-finding, placebo-controlled study in patients with chronic HIV infection and inadequate immune restoration treated with long-term highly active antiretroviral therapy (HAART). A total of 150 eligible subjects will be selected and randomized at a ratio of 1:1:1 into T8 0.5 mg QD, 1 mg QD, and placebo group, with background HAART unchanged, for 48 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese subjects aged 18-65, male or female；
2. Subjects with Body mass index (BMI) ≥18 (kg/m2); Male weight ≥50kg, female weight ≥45kg；
3. Subjects must meet the criteria;
4. No birth planning；
5. Understand and sign informed consent form voluntarily.

Exclusion Criteria:

1. allergic constitution；
2. Pregnant or lactating women；
3. Subjects who have been diagnosed with malignant tumors；
4. Subjects whose laboratory tests meet the conditions；
5. Subjects who have been diagnosed with severe gastrointestinal diseases；
6. Subjects who have been diagnosed with severe cardiovascular disease；
7. Subjects who have been diagnosed with severe cerebrovascular disease；
8. Subjects with history of alcohol and drug abuse；
9. Subjects who have participated in any other clinical trial；
10. Subjects who have any conditions that the investigator considers not suitable for this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
CD4+ T lymphocyte count | 48 week
  The changes of CD4+ T lymphocyte count from baseline
The proportion of subjects whose CD4+ T lymphocyte count increased by≥50 /μL from baseline | 48 week
  The proportion of subjects whose CD4+ T lymphocyte count increased by≥50 /μL from baseline
The changes of inflammatory factors | 48 week
  The quantitative changes of inflammatory factors（IP-10、hsCRP、IL-6）from baseline

SECONDARY OUTCOMES:
CD4+/CD8+T lymphocyte ratio | 24 week and 48 week
  The changes of CD4+/CD8+T lymphocytes from baseline
The proportion of subjects whose CD4+ T lymphocyte count is increased by ≥20% from baseline | 24 week and 48 week
  The proportion of subjects whose CD4+ T lymphocyte count is increased by ≥20% from baseline
The proportion of subjects whose CD4+ T lymphocyte count ≥ 200 /μL | 24 week and 48 week
  The proportion of subjects whose CD4+ T lymphocyte count after treatment is≥200/μL, among subjects with CD4+T lymphocyte counts < 200/μL at baseline.
Incidence of AE and SAE | 24 week and 48 week
  The incidence of AE and SAE

OTHER OUTCOMES:
The changes of the proportion of CD8+ T lymphocyte activation | 24 week and 48 week
  The changes of the proportion of CD8+ T lymphocyte activation (CD8+CD38+%，CD8+HLA-DR+%) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Taisheng Li, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Dita Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing You An Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Changsha, Changsha, Hunan
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Yun Provincial Infectious Disease Hospital, Kunming, Yunnan
  - Xixi Hospital of Hangzhou, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Tianjin Second People's Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cao W, Liu X, Han Y, Song X, Lu L, Li X, Lin L, Sun L, Liu A, Zhao H, Han N, Wei H, Cheng J, Zhu B, Wang M, Li Y, Ma P, Gao L, Wang X, Yu J, Zhu T, Routy JP, Zuo M, Li T. (5R)-5-hydroxytriptolide for HIV immunological non-responders receiving ART: a randomized, double-blinded, placebo-controlled phase II study. Lancet Reg Health West Pac. 2023 Mar 15;34:100724. doi: 10.1016/j.lanwpc.2023.100724. eCollection 2023 May. PMID 37283977